

# #2001957718 - Medication Adherence Given Individual SystemCHANGE(TM) in Advancing Nephropathy (MAGICIAN) Pilot Study

#### **Protocol Information**

| Review Type Expedited | Status Approved | Approval Date Oct 31, 2023 | Continuing Review Date Apr 09, 2020 |
|---|---|---|---|
| Expiration Date | Initial Approval Date Apr 09, 2020 | Initial Review Type Expedited | |

#### Feedback

| Approva <sup>I C</sup> ommen <sup>t</sup> |
|---------------------------------------------------------------------|
| <sup>A</sup> men <sup>d</sup> ment A016 |
| This research is approved under the following expedited categories: |
| _ Category 5 |
| _ Category 6 |
| _ Category 7 |

# **Protocol Amendment Form**

**Amendment Request** 

4000

### **Select your Protocol Type**

Expedited/Full Board

4012

#### **Amendment Number**

A016

4001

### Select the types of changes being made.

Other changes

4003

# Select the appropriate status of the study.

Closed to Enrollment – Research interventions continue

4004

# Describe the changes being made.

Those currently participating in the control intervention will be recruited to participate in the SystemCHANGE Intervention. IFC updated to reflect this change.

4005

# Why are these changes being made (i.e. what is the rationale for these changes)?

To increase understanding of how SystemCHANGE can increase medication adherence in those who have chronic kidney disease. Previous enrollment numbers are not significant for complete data analysis. Even though not a true crossover design, the increased enrollment in the SYstemCHANGE intervention will lead to better discoveries to yield R01 funding.

4006

# Will any previously enrolled subjects be informed of these changes?

No

4011

| <b>Expl</b> | lain | why | subj | jects | will | not | be | informed | d. |
|-------------|------|-----|------|-------|------|-----|----|----------|----|
|-------------|------|-----|------|-------|------|-----|----|----------|----|

Only those currently enrolled in the Main Study Control Intervention will be made aware of these changes and re-consented. Others who have completed the study will not be eligible for this change.

#### **General Information**

# **Principal Investigator**

Ellis, Rebecca

### Lead Unit

IN-NURS - NURSING

#### **Protocol Title**

Medication Adherence Given Individual SystemCHANGE(TM) in Advancing Nephropathy (MAGICIAN) Pilot Study

#### Personnel

Person

Ellis, Rebecca

Email Address

rjbartle@iu.edu

Researcher Role

Principal Investigator (PI)

| Home Unit |
|---|
| IN-NURS - NURSING |
| Contact Roles |
| Permissions |
| Full Access |
| Affiliation Type |
| Training |
| Behavioral/Social Science Researcher - Stage 1 - CITI 01/30/23 - 01/30/28 Biomedical Researcher - Stage 2 - CITI 09/19/22 - 09/18/27 |
| COI Disclosure Status: Approved Personnel Attachments |
| Person Hill, James |
| Tim, Garries |
| Email Address |
| hilljh@iupui.edu |
| Researcher Role |
| Key Personnel |
| Contact Roles |

| Permissions |
|---------------------------------------------------------------------------|
| Read-Only |
| Affiliation Type |
| IU |
| Training |
| Behavioral/Social Science Researcher - Stage 1 - CITI 10/13/20 - 10/12/25 |
| COI Disclosure Status: Approved |
| Personnel Attachments |
| r croomier Actuorimento |
| Person |
| Kerley, Denise |
| Email Address |
| kdkerley@iu.edu |
| Researcher Role |
| Key Personnel |
| Contact Roles |
| Contact Roles |
| Permissions |
| Read-Only |
| Affiliation Type |
| IU |

# Training Behavioral/Social Science Researcher - Stage 1 -Biomedical Researcher - Stage 1 - CITI 02/22/17 - 02/22/20 03/25/20 - 03/24/23 Expired Expired **COI Disclosure** Status: Approved Personnel Attachments Attachment $Kerley\_2020\_citiCompletionReport1927386.pdf$ Name Citi **Attachment Type** Other Comments Attachment Kerley\_032420\_updated Conflict Of Interest.pdf Name COL **Attachment Type** Site Specific Personnel List Comments

| Person | |
|---|---|
| Perkins, Susan | |
| Email Address | |
| sperkin1@iu.edu | |
| Researcher Role | |
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Read-Only | |
| Affiliation Type | |
| IU | |
| Training | |
| Biomedical Researcher - Stage 1 - CITI<br>09/27/22 - 09/26/27 | Behavioral/Social Science Researcher - Stage 4 -<br>CITI<br>09/27/22 - 09/26/27 |
| COI Disclosure | |
| Status: Approved | |
| Personnel Attachments | |
| Person | |
| Russell, Cynthia | |
| Email Address | |
| russellc@umkc.edu | |

| I |
|---|
| Researcher Role |
| Key Personnel |
| Contact Roles |
| Permissions |
| Affiliation Type |
| Non-Affiliated |
| Training Ourses on file. |
| COI Disclosure Status: Not Disclosed |
| Personnel Attachments |
| Personnel Attachments |
| Personnel Attachments Attachment |
| Personnel Attachments |
| Personnel Attachments Attachment |
| Personnel Attachments Attachment 1R21NR019348-01.pdf |
| Personnel Attachments Attachment 1R21NR019348-01.pdf Name Summary Statement |
| Attachment 1R21NR019348-01.pdf Name Summary Statement Attachment Type |
| Personnel Attachments Attachment 1R21NR019348-01.pdf Name Summary Statement |
| Personnel Attachments Attachment 1R21NR019348-01.pdf Name Summary Statement Attachment Type |
| Attachment 1R21NR019348-01.pdf Name Summary Statement Attachment Type Other |
| Attachment 1R21NR019348-01.pdf Name Summary Statement Attachment Type Other |

| Email Address | |
|----------------------------------------|----------------------------------|
| adsinha@iu.edu | |
| Researcher Role | |
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Read-Only | |
| Affiliation Type | |
| IU | |
| Training | |
| Biomedical Researcher - Stage 1 - CITI | VA Training - CITI |
| 11/15/22 - 11/15/27 | 11/17/17 - 11/17/21 (1) Expired |
| COI Disclosure<br>Status: Approved | |
| Personnel Attachments | |
| Person | |
| Zvonar, Sarah | |
| Email Address | |
| szvonar@iu.edu | |
| Researcher Role | |
| Key Personnel | |
| I . | |

| Contact Roles |
|---|
| Permissions |
| Full Access |
| Affiliation Type |
| IU |
| Training |
| Behavioral/Social Science Researcher - Stage 4 - CITI 08/31/21 - 08/30/26 |
| · |
| COI Disclosure<br>Status: Approved |
| Personnel Attachments |
| Person |
| Person Elomba, Charles |
| Elomba, Charles |
| Elomba, Charles Email Address |
| Elomba, Charles Email Address chelomba@iu.edu |
| Elomba, Charles Email Address chelomba@iu.edu Researcher Role |
| Elomba, Charles Email Address chelomba@iu.edu Researcher Role Key Personnel |
| Elomba, Charles Email Address chelomba@iu.edu Researcher Role Key Personnel |
| Elomba, Charles Email Address chelomba@iu.edu Researcher Role Key Personnel Contact Roles |
| Elomba, Charles Email Address chelomba@iu.edu Researcher Role Key Personnel Contact Roles Permissions |

| Affiliation Type | |
|---|---|
| IU | |
| Training | |
| Behavioral/Social Science Researcher - Stage 1 - CITI 05/16/22 - 05/15/27 | Biomedical Researcher - Stage 1 - CITI<br>05/07/22 - 05/06/27 |
| COI Disclosure Status: Approved Personnel Attachments | |
| Person | |
| Hays, Matthew | |
| Email Address | |
| maedhays@iupui.edu | |
| Researcher Role | |
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Read-Only | |
| Affiliation Type | |
| IU | |

# Training Behavioral/Social Science Researcher - Stage 1 -Biomedical Researcher - Stage 1 - CITI 09/13/21 - 09/12/26 09/13/21 - 09/12/26 Biomedical Researcher - Stage 2 - CITI 08/30/21 - 08/29/26 **COI Disclosure** Status: Approved Personnel Attachments Person Lillie, Matthew **Email Address** malillie@iu.edu Researcher Role Other Research Staff **Contact Roles Permissions** Read-Only **Affiliation Type** IU

#### **Training**

Behavioral/Social Science Researcher - Stage 1 - CITI

09/10/21 - 09/09/26

Biomedical Researcher - Stage 1 - CITI 09/10/21 - 09/09/26

COI Disclosure Status: Not Disclosed Personnel Attachments Person Carpenter, Janet **Email Address** carpentj@iu.edu Researcher Role Key Personnel **Contact Roles** Permissions Read-Only **Affiliation Type** IU Training Behavioral/Social Science Researcher - Stage 1 -Biomedical Researcher - Stage 1 - CITI CITI 05/06/22 - 05/05/27 08/27/10 - 08/26/13 Expired **COI Disclosure** Status: Approved Personnel Attachments

| Person |
|---------------------------------------------------------------------------|
| Draucker, Claire |
| Email Address |
| cdraucke@iu.edu |
| Caraucke@id.edd |
| Researcher Role |
| Key Personnel |
| Contact Roles |
| Contact Roles |
| Permissions |
| Read-Only |
| Affiliation Type |
| IU |
| Training |
| Behavioral/Social Science Researcher - Stage 4 - CITI 12/18/20 - 12/17/25 |
| COI Disclosure |
| Status: Approved |
| Personnel Attachments |
| Person |
| Short, Danielle |
| Email Address |
| shortdn@iu.edu |

| Researcher Role | |
|---|---|
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Read-Only | |
| Affiliation Type | |
| IU | |
| Training | |
| Behavioral/Social Science Researcher - Stage 1 - CITI 09/06/19 - 09/05/22 • Expired | Biomedical Researcher - Stage 1 - CITI<br>05/11/21 - 05/10/26 |
| COI Disclosure<br>Status: Expired | |
| Personnel Attachments | |
| Person | |
| Wilson, Sylvia | |
| Email Address | |
| sylwilso@iu.edu | |
| Researcher Role | |
| Key Personnel | |
| Contact Roles | |

| Permissions |
|---------------------------------------------------------------------------|
| Read-Only |
| Affiliation Type |
| IU |
| Troining |
| Training |
| Behavioral/Social Science Researcher - Stage 1 - CITI 06/04/22 - 06/03/27 |
| COI Disclosure |
| Status: Expired |
| Personnel Attachments |
| Person |
| Heck, Rachel |
| Email Address |
| reheck@iupui.edu |
| Researcher Role Koy Dorooppol |
| Key Personnel |
| Contact Roles |
| Permissions |
| Read-Only |
| Affiliation Type |
| IU |



| Person |
|---------------------------------------------------------------------------|
| Williams, Alexis |
| Email Address |
| aljewill@iu.edu |
| Researcher Role |
| Key Personnel |
| Contact Roles |
| Permissions |
| Read-Only |
| Read-Offiy |
| Affiliation Type |
| IU |
| Training |
| Behavioral/Social Science Researcher - Stage 1 - CITI 06/16/22 - 06/15/27 |
| COI Disclosure Status: Expired |
| Personnel Attachments |
| reisonnei Attachments |
| Person |
| Vires, Mandy |
| Email Address |
| mjvires@iu.edu |

| Researcher Role | |
|---|---|
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Read-Only | |
| Affiliation Type | |
| IU | |
| Training | |
| Behavioral/Social Science Researcher - Stage 1 - CITI 06/29/22 - 06/28/27 | |
| COI Disclosure Status: Expired | |
| Personnel Attachments | |
| | = |
| Person | _ |
| Person<br>Kerley, Basia | |
| Kerley, Basia | |
| Kerley, Basia Email Address | |
| Kerley, Basia Email Address bekerley@iu.edu | |
| Kerley, Basia Email Address bekerley@iu.edu Researcher Role | |
| Kerley, Basia Email Address bekerley@iu.edu Researcher Role Key Personnel | |
| Kerley, Basia Email Address bekerley@iu.edu Researcher Role Key Personnel | |

| Permissions | |
|---|---|
| Read-Only | |
| Affiliation Type | |
| IU | |
| Training | |
| Behavioral/Social Science Researcher - Stage 1 -<br>CITI<br>09/03/22 - 09/02/27 | Biomedical Researcher - Stage 1 - CITI 02/18/20 - 02/17/23 • Expired |
| COI Disclosure Status: Approved Personnel Attachments | |
| Person | |
| Elliott, Shannon | |
| Email Address | |
| sdelliot@iu.edu | |
| Researcher Role | |
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Read-Only | |
| Affiliation Type | |
| IU | |

| Training | |
|---|---|
| Behavioral/Social Science Researcher - Stage 1 - CITI 09/19/22 - 09/18/27 | Biomedical Researcher - Stage 1 - CITI<br>09/19/22 - 09/18/27 |
| COI Disclosure<br>Status: Approved | |
| ersonnel Attachments | |
| Person | |
| Miller, Courtney | |
| Email Address | |
| cousmill@iu.edu | |
| Researcher Role | |
| Key Personnel | |
| Contact Roles | |
| Permissions | |
| Affiliation Type | |
| IU | |
| Training | |

| Person |
|---------------------------------------------------------------------------|
| Bustin, Rebecca |
| Email Address |
| rbustin@iu.edu |
| Researcher Role |
| Key Personnel |
| Contact Roles |
| Permissions |
| Read-Only |
| Affiliation Type |
| IU |
| Training |
| Behavioral/Social Science Researcher - Stage 1 - CITI 01/27/23 - 01/27/28 |
| COI Disclosure |
| Status: Approved |
| Personnel Attachments |
| Person |
| Kapunan, Andrei |
| Naparian, Anarei |
| Email Address |
| akapunan@iu.edu |

| Researcher Role |
|---|
| Key Personnel |
| Contact Roles |
| Permissions |
| Read-Only |
| Affiliation Type |
| IU |
| Training |
| Behavioral/Social Science Researcher - Stage 1 - CITI 02/26/23 - 02/26/28 |
| COI Disclosure<br>Status: Approved |
| Status. Approved |
| Personnel Attachments |
| Personnel Attachments |
| Personnel Attachments Person |
| Personnel Attachments Person Hoffman, Colin |
| Personnel Attachments Person Hoffman, Colin Email Address |
| Personnel Attachments Person Hoffman, Colin Email Address cwhoffma@iu.edu |
| Person Hoffman, Colin Email Address cwhoffma@iu.edu Researcher Role Key Personnel |
| Personnel Attachments Person Hoffman, Colin Email Address cwhoffma@iu.edu Researcher Role |
| Person Hoffman, Colin Email Address cwhoffma@iu.edu Researcher Role Key Personnel |

| | Permissions |
|---|------------------------------------------------------------|
| | Read-Only |
| | Affiliation Type |
| | IU |
| | Training |
| | Biomedical Researcher - Stage 1 - CITI 08/03/22 - 08/02/27 |
| | COI Disclosure<br>Status: Approved |
| F | Personnel Attachments |
| | Protocol Type |
| | Select Protocol Type Expedited |
| | Participant Type |
| | Participant Information |
| | Participant Type |
| | Total |
| | Participant Number 150 |

**Organizations Organizations List** Organization **IU HEALTH** Organization **ESKENAZI HEALTH** Organization INDIANA UNIVERSITY (UA) **Funding** Will the study be funded, fully or partly by, any of the following sources (this includes pass through funding)? Select all that apply. Federal funding **Funding Sources Funding Source** NATIONAL INSTITUTE OF NURSING RESEARCH

**Conflicts of Interest** 

Are any of the investigators listed in the personnel section aware of an institutional conflict of interest which could affect or be affected by this research?

No

q24901

Do any of the investigators listed in the Personnel section (or their immediate family members) have a significant financial interest which could affect this research?

No

q24905

Does the Principal Investigator affirm all investigators listed as personnel on this protocol have agreed to participate in this project, are aware of their status and role, and have been adequately trained to participate in the project?

Yes

**A-Level of Review** 

q720

Does any research activity in this study present more than minimal risk to human subjects?

No. The research may qualify for Expedited review if all research procedures fall into one of the categories below.

## Check all category(ies) which apply to this research.

Category 5 - Research involving materials (data, documents, records, or specimens) that have been collected, or will be collected solely for nonresearch purposes

Category 6 - Collection of data from voice, video, digital or image recordings made for research purposes

Category 7 - Research on individual or group characteristics or behavior, or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies

q724

Will the researchers be using a data collection form? Yes. It is/will be attached.

q23340

Would identification of subjects and/or their responses reasonably place them at risk for any of the following (check any that apply):

None

**B-Lay Summary Research Design** 

# Describe the purpose of this study in lay terms, including research question(s) and hypothesis.

The purpose of this-group, randomized, controlled trial is to evaluate the refined SystemCHANGE™ against attention control patient education in CKD patients taking RAAS medications. Patients will be recruited from two sources: 1) the largest and most comprehensive health care system in the state and 2) one of the largest essential health care systems in the country. Data are collected at baseline, 8 weeks(immediately post-intervention) and 12 weeks. Specific aims are to: Aim 1. Estimate acceptability, outcome expectancy and credibility of the refined SystemCHANGE™ Intervention and for the attention control at 8 and 12 weeks after baseline. Aim 2. Estimate preliminary efficacy of SystemCHANGE™ Intervention versus attention control on medication adherence (primary outcome) and personal systems behavior (mechanism of action) at 8 and 12 weeks among people with CKD taking a once-daily RAAS inhibiting medication. The immediate impact of this study will be data to inform the design of a future, fully powered, efficacy trial. If findings are as expected, we will proceed to an R01 application. If findings are not as expected (e.g., negative), we will work to improve the SystemCHANGE™ intervention or move to a different intervention in future trials. The long-term impact of this line of research will be additional empirical evidence for novel medication adherence interventions in this population to inform future evidence-based guidelines, position statements, and practice recommendations.

List and describe all research interactions and/or interventions, including the frequency and duration of procedures, and length of participation for individual subjects.

WHAT WILL HAPPEN DURING THE STUDY? This study has 3 phases-the screening phase, the intervention phase, and the maintenance phase. Before being invited to participate in this study, you will be asked questions from the 6-item cognitive screening survey to make sure you qualify for the study. Screening Phase If you are eligible to take part in the study, we will begin by reviewing your medical records for medications you take, what level of renal impairment you have, and may periodically review your records if you have medication changes or visits with your doctor or hospital. After this review, with the study nurse, we will ask you to fill out a demographics form. After this, we will monitor how you take your medication by giving you a pill bottle to use that has an electronic cap that will let us know when and how often you open the pill bottle to take a pill. For two months, you will use this special pill bottle and remove the cap when you normally take your medication. After you take your medication, you will put the cap back on the bottle. You will also be given a discrepancy log to make notes on your medication taking. The first and the fourth week the study nurse will call you to ask how you are using the pill bottle and cap to make sure you are not having any problems using it. At the end of the two-months, someone from our study team will call you and tell you how to mail the empty bottle and cap back to the study team. At this time, we will ask you survey questions about using the Mems and the patient activation measure (PAM-13). The study team will give you a pre-paid envelope to return the bottle and cap. Then you can mail it back to us by putting the sealed envelope in a US postal mailbox. The study investigator will then look at the information from the cap and if you have a medication score of less than 0.85, we will ask you to continue in the study. If your score is 0.85 or greater, we will thank you for your participation and you will end the study. If you are invited to participate in the next phase of the study, we will randomly assign you to treatment group 1 or treatment group 2. Random assignment is like flipping coin-heads put you in one group and tails puts you in the other group. Both groups will get an intervention for improving kidney health. Intervention Phase The intervention phase is next. If you are invited to continue the study, we will arrange a time to contact you via telephone or

virtually. Before that meeting, your electronic cap, and the bottle will be returned to you and you will be asked to use it for 12 more weeks. You will also be asked to complete additional surveys. These surveys include 1) Acceptability Scale, 2) Outcome Expectancy, 3) Treatment Credibility Questionnaire. You will again use a special bottle and cap to keep and take your medication. You will also be given a special mobile phone for this study. Each week for 6 weeks, you will place the phone near the bottle to send data to the study team. After the data is received, you will get one text message on the provided mobile phone each week for 6 weeks. These text messages are education about your disease and disease process. A member of our study team will call you each week to ask you questions and make sure the equipment is working correctly. The study team member will also discuss information from the first visit with you. We will also ask you about any healthcare visits that you have with your healthcare provider. This might include a visit to your providers for a checkup and any time spent in the hospital or a visit to the emergency room. Treatment group 1 will receive education that will help to learn more about caring for your chronic kidney disease. You will receive your first materials during the research nurse's visit to your home. You will receive a telephone call from the research nurse to review and discuss the educational materials throughout the study. In addition, the research nurse will ask you if you have had any changes to your medications and what healthcare providers you have seen recently. Treatment group 2 will receive training by a research nurse who will work with you to learn about SystemCHANGE™. You will get a printer report from the MEMS cap to see how you are doing with taking your medications. Part of this intervention involves completing time worksheets together with the study nurse (Important People Form, Life Routine Form, Solutions Form). This helps you identify people who are important in helping you with taking your medicines, and identify your daily routines, specifically the routines around the times that you are scheduled to take your medicines. The research nurse will ask you to think about possible changes in your routines that may make it easier for you to take your medicines every day on time without having to remember. The research nurse will call you to discuss the important people you marked on the Important People Form and which solutions you have decided to use from the Solution Form. Throughout the study, the research nurse will send your personal medication-taking report. The research nurse will then telephone you to discuss how you are doing with taking your medicine every day on time using the forms. Together, you will discuss

possible solutions for improving your medication taking. You will try out the ideas and then see if your medication-taking is getting better from your personal medication-taking report. In addition, the research nurse will ask you if you have had any changes to your medications and what healthcare providers you have seen. Amended procedures. We are inviting participants who have completed Treatment group 1 to complete Treatment Group 2 intervention as well. Participation in this additional study of Treatment group is voluntary. If you chose to also participate in Treatment Group 2, you will follow the procedures outlined above, starting with the intervention phase after you have consented to participate. You will be asked to keep using the electronic pill bottle for 12 more weeks. You will also be asked to complete additional surveys. These surveys include 1) Acceptability Scale, 2) Outcome Expectancy, 3) Treatment Credibility Questionnaire. You will keep using the special mobile phone for this study. Each week for 6 weeks, you will place the phone near the bottle to send data to the study team, like you have been doing. After the data is received, you will get one text message on the provided mobile phone each week for 6 weeks. These text messages are education about your disease and disease process. A member of our study team will call you each week to ask you questions and make sure the equipment is working correctly. The study team member will also discuss information from the first visit with you. We will also ask you about any healthcare visits that you have with your healthcare provider. This might include a visit to your providers for a checkup and any time spent in the hospital or a visit to the emergency room. The group who has completed Treatment group 1 will follow the protocol for Treatment group 2. Participants will receive training by a research nurse who will work with you to learn about SystemCHANGE™. Part of this intervention involves completing time worksheets together with the study nurse (Important People Form, Life Routine Form, Solutions Form). This helps you identify people who are important in helping you with taking your medicines, and identify your daily routines, specifically the routines around the times that you are scheduled to take your medicines. The research nurse will ask you to think about possible changes in your routines that may make it easier for you to take your medicines every day on time without having to remember. The research nurse will call you to discuss the important people you marked on the Important People Form and which solutions you have decided to use from the Solution Form. Throughout the study, the research nurse will send your personal medication taking report to your phone. The research nurse will telephone you

to discuss how you are doing with taking your medicine. Together, you will discuss possible solutions for improving your medication taking. You will try out the ideas and then see if your medication taking is getting better from your personal medication taking report. In addition, the research nurse will ask you if you have had any changes to your medications and what healthcare providers you have seen. Maintenance Phase In both groups, at 6 weeks, someone from the study staff will call you and ask you some of the same questions as before about your medication and your kidney health, as well as repeat the previous surveys. They will also ask you some questions about participating in the study. In this final phase, you will continue to use the electronic cap and bottle to take your medications. At the end of the twelve weeks, you will once again take the surveys as before. You will receive a postage-paid envelope to return the cap to the study nurse. At this time, you will also take part in a semi-structured interview. In both groups, all of the interactions that you have with the study nurse over the telephone and virtually will be audiotaped so that the investigator can make sure the study nurse is following the research study steps. At the completion of the twelve weeks, you will have no additional testing in the study and you will continue to follow-up with your providers.

q23358

Will any non-English study documents be uploaded?

q24919

Is this research funded by, or has a funding application been submitted to, a federal agency? This includes federal passthrough funding.

Yes

q25019

. P<sub>rov</sub>id<sub>e t</sub>he name of the federal funding agency



### List inclusion criteria - eligibility criteria for subjects.

(1) age > 18 years, (2) prescribed at least 1 daily RAAS inhibiting medication, (3) CKD diagnosis eGFR category G1 to G4, (4) RAAS inhibiting medication adherence of <.85 documented during screening (5) proteinuria defined as a urine Protein-to-Creatinine ratio > 150 mg/g or urine Albumin-to-Creatinine ratio >30mg/g (6) able to speak, hear, and understand English determined by the ability to participate and comprehend conversation about potential inclusion in the study, (7) self-reported ability to open a pill cap, (8) able to self-administer RAAS inhibiting medications, (9) willing to use a study phone, (10) has no cognitive impairment as determined by a score of 4 or greater on the 6-item Telephone Mental Status Screen Derived from the Mini-Mental Status Exam73 (cognitive screener), (11) has no other diagnoses that may shorten life span, such as metastatic cancer, (12) is not hospitalized, (13) receives care through IUH or Eskenazi.

q23235

# List exclusion criteria (any criteria which would exclude otherwise acceptable subjects).

Participants with kidney failure defined by GFR <15 mL/min/1.73m2.13 Participants will be excluded if they are receiving dialysis or have dialysis access placed (e.g., graft or arteriovenous fistula) in anticipation of starting dialysis. Kidney and kidney-pancreas transplant recipients will be excluded. Participants will be excluded if they have another medication adherence strategy in place (e.g., medication adherence pill packs or blister packs from a pharmacy).

Will subjects be paid for their participation in the study? Payment includes reimbursement of expenses (other than compensation for injury).

Yes

q23347b

# Describe the payment arrangement, including amount and timing of disbursement.

Participants will be paid \$20 honorarium at screening completion. We will pay participants in the intervention and attention control groups \$30 at the study end to thank them for their time. For those who participate in both treatment groups. As a thank you, you will receive \$30 at the completion of the 12-week educational intervention as well as \$30 at the completion of the 12-week SystemCHANGE™ intervention. This will be mailed to you within 10 days of receipt of the study materials.

q23348

Justify the proposed payment arrangement described above, specifically why payment does not provide undue influence for subject participation.

The amount recognizes the commitment time by the participant, yet a relatively minimal amount that is consistent with other behavioral studies.

q23349

Will partial payment be provided if the subject withdraws prior to completion of the study?

No

# Explain why failure to offer partial payment will not unduly influence subjects to complete the study.

Payments are associated with specific phases of the study and a minimal amount, and providing partial payments would not reflect positively to patient participants. Payment compensations are provided after each phase.

q23352

# Does this research involve (choose all that apply):

- the STUDY of any of the following products (regardless of FDA approval status). "The study of" means at least one objective of the study is related to obtaining data about the product
- USE of any of the following products which have not been cleared or approved by the FDA for use in the US
- USE of any of the following products for open label extension, treatment, or compassionate use

NONE

q23454a

## This research involves (check all that apply):

None of the Above

q25049a

### Is this research considered a prospective clinical study?

Yes - This study may require entry in OnCore.

q30000a

### Is this community-engaged research?

No

**C-Sites and Collaborations** 

| q700 |
|---|
| Are there additional locations of research, not already listed? No |
| q704 |
| Are you requesting that IU provide IRB approval for any researchers who are NOT IU affiliates? No |
| q710a |
| Is this a multi-center study or multi-site clinical trial? No |
| D-Recruitment Methods |
### Describe how potential subjects will be initially identified.

There will be multiple forms of recruitment. Eligible patients will be identified by Regenstrief recruitment core based on inclusion criteria. Co-I Sinha will obtain permission from nephrology colleagues through IUHP for permission to contact their patients using an opt-out recruitment strategy with letters mailed to eligible individuals home address. Letters will be mailed to eligible patients introducing the opportunity to participate in the study. Patients who wish to opt-out or opt-in do so by contacting the phone number identified on the recruitment materials and/or following the instructions on the mailed letter. After these letters are mailed, participants will be contacted in randomized order from this Regenstrief list of potential participants. In addition to the self-referral, opt-out procedures, and phone calls from the Regenstrief list; participants will be recruited in the clinics in a face-to-face fashion. Physicians and staff will identify potential participants, with the help of the research assistant, and ask potential participants if they would be willing to speak with the research assistants about potential involvement. Research assistants present in the clinic will be wearing attached buttons.

q30002

## Check any of the following sources of information which will be used to identify potential subjects.

Subject self-referral in response to recruitment materials Medical records or clinic schedules Physician/provider referral Other

q30002C5Text

## Explain the Other source(s) of information which will be used to identify potential subjects.

Regenstrief Data Core Clinic Schedules Medical Records

### Describe how potential subjects will be initially contacted.

Regenstrief will generate a patient list. The resulting list of patients will be used as a sampling pool. Using a computer-generated list of random numbers the biostatistician produces, the RA will randomly select each potential subject from the list. The RA will contact identified patients and ask if they are willing to discuss possible participation in a study. Brochures will be utilized to introduce the participants briefly to the study and introduce them to the study team. Participants will be identified prior to their scheduled clinic visit from clinic schedules then verified with medical records for inclusion and exclusion criteria. Flyers in the patient facing areas will give general information about qualifications and process of the MAGICIAN study, as well as information to contact MAGICIAN team. A physician and staff flyer will give general information for the staff if general questions are asked when a research assistant is not present or with another potential participant.

q23237

## Check any of the following recruitment materials which will be used to contact potential subjects.

Direct Mail/Email Flyers/Brochures Verbal Scripts

q25426b

### Select any of the following circumstances which apply to this research.

None of the above.

q23245

Would participation in this study preclude subjects from participating in other research studies?

No

q23296

List and describe (in lay terms) the potential risks to which subjects may be exposed as a result of their participation in the research.

While participating in the study, the risks, side effects, and/or discomforts include: • Possible frustration when using the electronic medication monitoring (EMM) cap • Fatigue (physical or mental during answering the questions • Possible loss of confidentiality • Uncomfortable answering personal questions

q23297

Describe procedures for protecting against, or minimizing, the potential risks listed above. Include any procedures that are already being performed on subjects for diagnostic, treatment, or standard purposes.

We will minimize these risks by: • Hiring Research Assistants and Nurse Intervenors who have education and experience working with people with health conditions • Making sure you are comfortable using the EEM cap before starting this study and checking on you weekly for issues. • To minimize possible fatigue, you will be asked every 20 minutes during the interviews if you would like to take a break. • Keeping all files in a locked, secure, location available only to the research team. • If uncomfortable with questions, tell the researcher you do not want to answer that particular question • Face-to-face recruitment will be in an area away from the other patients and staff in the clinic setting.

# Explain how research data will be protected so that only approved persons have access to subjects' identifiable data (i.e. confidentiality of data).

The PI will be responsible for all data management. Study participants' (Pps) confidentiality will be maintained using the following techniques: (1) each Pp will be given a unique study identification code to enable data source merging, e.g. demographics, MEMs Capmedication adherence data, (2) the unique study identification codes will be stored in a locked separate file, (3) all electronic data will be stored in password-protected files, in password-protected computers. All data hard copies will be stored in the PIs' locked office, in locked file cabinets, and (4) all Pp names and other identifiers will be removed from the data upon assignment of a study identification code

q23300

# Explain how subjects' physical privacy will be protected, both during recruitment/screening and during participation in the research.

The patients' physical privacy will be maintained by recruitment materials sent to possible participants' homes. Potential participants arriving in the clinic will interact with the research staff in a private area with MAGICIAN research assistants who have passed required CITI training as well as background checks. Interviews throughout the study are conducted via phone or virtually. Interactions of text messages and phone calls will be during the participants choosing.

q23301

Is there a potential for subjects to benefit directly from participation in the study?

Yes

q23302

# Describe the potential benefits to be gained by the individual SUBJECT. Please note that payment for participation is not considered a benefit.

As a result of this study, we anticipate that the participants may take their medications better, contributing to better adherence.

q23303

## State the potential benefits or information which may accrue to SCIENCE or SOCIETY in general as a result of this work.

The immediate impact of this study will be data to inform the design of a future, fully powered, efficacy trial. If findings are as expected, we will proceed to an R01 application. If findings are not as expected (e.g., negative), we will work to improve the SystemCHANGE™ intervention or move to a different intervention in future trials. The long-term impact of this line of research will be additional empirical evidence for novel medication adherence interventions in this population to inform future evidence-based guidelines, position statements, and practice recommendations.

F-Data Safety Monitoring

q23304

Describe the provisions for monitoring the data to ensure the safety of subjects.

Complete plan in attachment.

**H-Informed Consent** 

Will all or some subjects consent to participate in the research?

All subjects (or their legally authorized representative) will consent to participate in the research

q909

For those subjects who will consent to participate, explain how subjects (or subjects' legally authorized representative) will be presented with the information needed to decide to participate, including all elements of informed consent.

Recruitment sites will generate lists of potentially eligible patients using electronic health record data to ensure a match with eligibility requirements with regard to prescribed RAAS inhibitors, diagnosis and stage of CKD and proteinuria. The study staff will randomly select each potential participant from the list using a biostatistician produced list of random numbers, and mail letters to identified patients describing the study and opt-out procedures to avoid being contacted by the study staff. The study staff will contact patients by phone to discuss possible study participation and, if interested, verify study eligibility including administering the cognitive screener. If interested and eligible, the study staff will mail consent documents with instructions for returning them by mail/email. After receiving the signed consent, the participant will move into the screening phase. Staff will record reasons for those not eligible or not interested in the study.

Describe any informed consent tools which will be used to present information to potential subjects (i.e. consent documents, videos, brochure, drug/device information, etc) and how they will be used.

Informed consent documents will be mailed to the participants and asked to be mailed back after the initial screening of inclusion/ exclusion criteria and an informal agreement to participate. The initial screening via telephone will provide details of the study including any risks or benefits as well as answer any questions pertaining to the study. The informed consent documents also provide an opt-out at any time by contacting the primary investigator (Rebecca Ellis) at (317)274-0047. In clinic recruitment participants will complete the informed consent at time of contact.

q925

Describe the timing of the informed consent process, including how you will ensure potential subjects have sufficient opportunity to discuss and consider participation before agreeing to participate in the research.

Because the initial screening takes place via telephone and informed consent is to be obtained via mail for participation, there is a period of days between the telephone call, returned signed consents, and an initial visit via phone or virtually. This ensures that participation is voluntary, there is sufficient time to consider participation, and multiple opportunities to discuss involvement further, as well as change their decision.

q30127a

Will you include all required elements of consent in your consent process?

Yes

Indicate in what language(s) the consent conversation will be conducted.

English

q926

Explain how you will ensure potential subjects understand the information you have presented to them before they agree to participate in the study.

We will leave time for questions with potential participants. We will utilize the "teach back" method to allow participants a chance to explain the information given to them about the study in their own terms.

q929

Briefly describe any training provided to investigators who are obtaining informed consent.

Staff will be trained rigorously in study procedures. Prior to the start of the study, staff will engage in role-play and simulation. All staff working on this study have completed CITI training.

q931

Does the research include any minimal risk procedures to which subjects will not consent?

No

q23678a

For those subjects who will consent to participate, choose whether the consent process will be documented by a written signature from subjects.

All consented subjects will provide a written signature as documentation of consent.

q30129a

Will subjects participate in any study activity prior to physically signing a consent document?

No

q940a

## Explain the process for obtaining a written signature from subjects.

After names are given by the provider, then randomly selected to be contacted for potential participation in this study, the participants are contacted via telephone for initial screening of inclusion/ exclusion criteria. The consent form is mailed to participants and the signed consent form will be mailed back with a provided self-addressed, stamped envelope before participation in this study. Those recruited in the clinic setting will be informed of the study procedures and two informed consents, one to sign and one to maintain for their records.

#### K-HIPAA

q23253

Are you part of a covered entity (health care provider that transmits health information electronically) or are you receiving information from a covered entity as part of your research?

Yes

q23254

Will protected health information be utilized, accessed, collected, or generated as part of the study?

Yes

q30347a

Select the electronic systems to be used for the collection and/or storage of protected health information (ePHI). Choose all that apply.

REDCap

q23257

Will you be accessing or collecting protected health information for RECRUITMENT purposes?

Yes

q23258

Choose all that apply to the recruitment plans.

Health information provided by clinicians not part of the study team

q23271

Will the clinician direct the potential subject to contact the study team?

Yes

q23277

HIPAA applies to your study, and requires that you obtain authorization for PARTICIPATION in research, or that you request a waiver. Check all that apply.

I will obtain written, signed authorization from subjects prior to their participation

q23278

Will you be collecting information from subjects' medical records?

Yes, I have uploaded an Authorization template to the Attachments section.

Attachment Type **Data Collection Instrument** Attachment EMM Discrepancy Log.docx Name **EMM Discrepancy Log** Comments Attachment Type Data Collection Instrument Attachment 13 Health Care Use Form Revision 3.docx Name Health Care Use, Medical Appointments Form Comments Attachment Type **Data Collection Instrument** Attachment

9BIntervention Steps 1 and 2 Important People Etc. Forms Revision 2.docx

| Name Important People Form, Life Routine Form, Solutions Form |
|---------------------------------------------------------------|
| Comments |
| Attachment Type |
| Data Collection Instrument |
| Attachment |
| 9C Intervention Steps 3 and 4 Questions.docx |
| Name |
| Questions for SystemCHANGE |
| Comments |
| Attachment Type |
| Data Collection Instrument |
| Attachment |
| PAM-13 .docx |
| Name |
| PAM-13 |
| Comments |
| Attachment Type Data Collection Instrument |

| Attachment |
|--------------------------------------------------|
| RO1_Ellis_Medical History.docx |
| Name |
| Medical Record Form |
| Comments |
| Attachment Type |
| Data Collection Instrument |
| Attachment |
| Social Support Appraisal.docx |
| Name |
| Social Support Appraisal |
| Comments |
| Attachment Type |
| Data Collection Instrument |
| Attachment |
| Acceptability Scales to add to appendix JSC.docx |
| Name |
| Acceptability Scale |
| Comments |

Attachment Type Data Collection Instrument Attachment R21\_Acceptability\_Scale (1).docx Name Accept Comments Attachment Type Data Collection Instrument Attachment EllisAppendix-3.pdf Name Mental Status Screen, Systems Thinking, Demographic Form, Electronic Medication Monitoring Discrepancy Log, Medical History data collection form questionnaire, Perceived Health Status Comments Attachment Type HIPAA Authorization Form Attachment MAGICIAN HIPPA.docx

| Name |
|---|
| HIPPA |
| Comments |
| Attachment Type |
| Protocol |
| Attachment |
| R21_MAGICIAN_Intervention Figure2 Updated.xlsx |
| Name |
| Figure 2 restart |
| Comments |
| Attachment Type |
| Attachment Type Recruitment Materials |
| Recruitment Materials |
| Recruitment Materials Attachment |
| Recruitment Materials Attachment Recruitment Script 10.31.2023.docx |
| Recruitment Materials Attachment Recruitment Script 10.31.2023.docx Name |
| Recruitment Materials Attachment Recruitment Script 10.31.2023.docx Name Script for phone calls |

| Attachment |
|----------------------------------------|
| Brochure MAGICIAN Final.pptx |
| Name |
| Brochure for participants |
| Comments |
| Attachment Type |
| Recruitment Materials |
| Attachment |
| Recruitment Letter Final- restart.docx |
| Name |
| Recruitment letter |
| Comments |
| Attachment Type |
| Recruitment Materials |
| Attachment |
| Amended_MAGICIAN_DSM.docx |
| Name |
| Comments |

| Attachment Type |
|--------------------------------------------|
| Recruitment Materials |
| Attachment |
| MAGICIAN_STUDY-physician flyer 7.11.22.png |
| Name |
| Comments |
| Confinents |
| Attachment Type |
| Recruitment Materials |
| Necruitment waterials |
| Attachment |
| Magician Patient Pamphlet copy.png |
| Name |
| Name |
| Comments |
| Attachment Type |
| Recruitment Materials |
| Attachment |
| KIDNEY DESIGN.pdf |
| NIBRET SEGION.pd. |
| Name |
| Comments |

т

| Attachment Type |
|---|
| Other |
| Attachment MAGICIAN IFC amended letter.docx |
| Name |
| Comments |
| Attachment Type |
| Recruitment Materials |
| Attachment MAGICIAN Study Image Flow _RJE.docx |
| Name |
| Imagery for recruiting to streamline conversations with potential participants. |
| Comments |
| Attachment Type |
| Recruitment Materials |
| Attachment Clinic RA Screening Tool.docx |
| Name |
| Screening tool to facilitate conversations between RA's and Physicians |

Г

٦

| Comments |
|--------------------------------------|
| Attachment Type |
| Informed Consent Statement |
| Attachment |
| Final _MAGICIAN_IFC_10.31.2023.docx |
| Name |
| Comments |
| End of Protocol Form KC IRB History |
| approvalDate |
| April 9, 2020 |
| FOR HSO OFFICE USE ONLY |
| Action History |
| Description |
| Expedited Approval |
| Date |
| Date January 8, 2021 |

Action Date January 8, 2021 Comments Amendment-004: Approved **Updated By** slbenken **Update Time** 2021-01-08T12:00:00.000Z Description Assigned to Agenda Date January 8, 2021 Action Date January 8, 2021 Comments Amendment-004: **Updated By** slbenken Update Time 2021-01-08T12:00:00.000Z Description

Submitted to IRB

Date January 6, 2021 **Action Date** January 6, 2021 Comments Amendment-004: Submitted to IRB **Updated By** rjbartle **Update Time** 2021-01-06T12:00:00.000Z Description Returned To PI Date December 8, 2020 **Action Date** December 8, 2020 Comments Amendment-004: Open for Incomplete Submission **Updated By** shream **Update Time** 2020-12-08T12:00:00.000Z

| Description |
|----------------------------------------------------------|
| Submitted to IRB |
| D. A. |
| Date December 7, 2020 |
| December 7, 2020 |
| Action Date |
| December 7, 2020 |
| 0.0000000000000000000000000000000000000 |
| Comments And any discount CO As Code resists of the IDD |
| Amendment-004: Submitted to IRB |
| Updated By |
| szvonar |
| Update Time |
| 2020-12-07T12:00:00.000Z |
| Description |
| Amendment Created |
| Date |
| December 7, 2020 |
| Action Date |
| December 7, 2020 |
| Comments |
| Amendment-004: Created |
| Updated By |
| szvonar |
| I |

Update Time

2020-12-07T12:00:00.000Z

Description

**Administrative Correction** 

Date

August 2, 2020

**Action Date** 

August 2, 2020

Comments

updating funding

Updated By

larcohen

Update Time

2020-08-02T12:00:00.000Z

Description

Amendment Deleted

Date

July 13, 2020

**Action Date** 

July 13, 2020

Comments

Amendment-003: Deleted - Delete amendment 3. (2001957718A003) I didn't realize Cynthia Russell was on there already. I do not have anything new to add.

**Updated By** 

szvonar

**Update Time** 

2020-07-13T12:00:00.000Z

Description

**Amendment Created** 

Date

July 13, 2020

**Action Date** 

July 13, 2020

Comments

Amendment-003: Created

**Updated By** 

szvonar

**Update Time** 

2020-07-13T12:00:00.000Z

Description

**Expedited Approval** 





Update Time
2020-07-13T12:00:00.000Z

Description

Submitted to IRB

Date

July 9, 2020

**Action Date** 

July 9, 2020

Comments

Amendment-002: Submitted to IRB

**Updated By** 

szvonar

**Update Time** 

2020-07-09T12:00:00.000Z

Description

Returned To PI

Date

July 6, 2020

**Action Date** 

July 6, 2020

Comments

Amendment-002: Open for Intake Pre-review

Updated By shream Update Time 2020-07-06T12:00:00.000Z Description Submitted to IRB Date July 2, 2020 **Action Date** July 2, 2020 Comments Amendment-002: Submitted to IRB Updated By szvonar Update Time 2020-07-02T12:00:00.000Z Description **Amendment Created** Date July 2, 2020 **Action Date** July 2, 2020

Comments Amendment-002: Created Updated By szvonar **Update Time** 2020-07-02T12:00:00.000Z Description **Expedited Approval** Date April 29, 2020 **Action Date** April 29, 2020 Comments Amendment-001: Approved Updated By pattonle Update Time 2020-04-29T12:00:00.000Z Description Assigned to Agenda

Date

April 29, 2020

Action Date April 29, 2020 Comments Amendment-001: **Updated By** pattonle **Update Time** 2020-04-29T12:00:00.000Z Description Submitted to IRB Date April 29, 2020 **Action Date** April 29, 2020 Comments Amendment-001: Submitted to IRB **Updated By** pattonle Update Time 2020-04-29T12:00:00.000Z Description

Returned To PI

| Date | |
|---|---|
| April 29, 2020 | |
| Action Date | |
| April 29, 2020 | |
| Comments Annual discount CO1: | |
| Amendment-001: | |
| Updated By | |
| pattonle | |
| Update Time | |
| 2020-04-29T12:00:00.000Z | |
| Description | |
| | - 1 |
| Submitted to IRB | |
| Submitted to IRB Date | |
| Date April 21, 2020 | |
| Date April 21, 2020 Action Date | |
| Date April 21, 2020 | |
| Date April 21, 2020 Action Date | |
| Date April 21, 2020 Action Date April 21, 2020 | |
| Date April 21, 2020 Action Date April 21, 2020 Comments Amendment-001: Submitted to IRB | |
| Date April 21, 2020 Action Date April 21, 2020 Comments | |
| Date April 21, 2020 Action Date April 21, 2020 Comments Amendment-001: Submitted to IRB Updated By | |
| Date April 21, 2020 Action Date April 21, 2020 Comments Amendment-001: Submitted to IRB Updated By | |

Description Returned To PI Date April 21, 2020 **Action Date** April 21, 2020 Comments Amendment-001: Open for Intake Pre-review Updated By shream Update Time 2020-04-21T12:00:00.000Z Description Submitted to IRB Date April 20, 2020 **Action Date** April 20, 2020 Comments Amendment-001: Submitted to IRB **Updated By** szvonar

Update Time 2020-04-20T12:00:00.000Z

Description

**Amendment Created** 

Date

April 20, 2020

**Action Date** 

April 20, 2020

Comments

Amendment-001: Created

**Updated By** 

szvonar

Update Time

2020-04-20T12:00:00.000Z

Description

**Expedited Approval** 

Date

April 9, 2020

**Action Date** 

April 9, 2020

Comments

Updated By pattonle Update Time 2020-04-09T12:00:00.000Z Description Assigned to Agenda Date April 9, 2020 **Action Date** April 9, 2020 Comments **Updated By** pattonle **Update Time** 2020-04-09T12:00:00.000Z Description Submitted to IRB Date April 9, 2020 **Action Date** April 9, 2020

| Comments |
|-----------------------------|
| Submitted to IRB |
| Updated By |
| pattonle |
| Update Time |
| 2020-04-09T12:00:00.000Z |
| Description Returned To PI |
| Returned to Pi |
| Date |
| April 9, 2020 |
| Astion Date |
| Action Date |
| April 9, 2020 |
| Comments |
| Updated By |
| pattonle |
| Update Time |
| 2020-04-09T12:00:00.000Z |
| Description |
| Submitted to IRB |
| Date |
| Date April 9, 2020 |
| April 8, 2020 |

| Action Date |
|--------------------------|
| April 8, 2020 |
| Comments |
| Submitted to IRB |
| Submitted to IND |
| Updated By |
| szvonar |
| Update Time |
| 2020-04-08T12:00:00.000Z |
| Description |
| Returned To PI |
| Date |
| April 6, 2020 |
| 7.p |
| Action Date |
| April 6, 2020 |
| Comments |
| Updated By |
| pattonle |
| Update Time |
| 2020-04-06T12:00:00.000Z |
| 2020 0 . 00 . 12.00.0002 |
| Description |

| I |
|---|
| Date |
| April 6, 2020 |
| Action Date |
| April 6, 2020 |
| Comments |
| Submitted to IRB |
| Submitted to IKD |
| Updated By |
| szvonar |
| Update Time |
| 2020-04-06T12:00:00.000Z |
| Description |
| Returned To PI |
| Returned To PI |
| Returned To PI Date |
| Returned To PI |
| Returned To PI Date March 30, 2020 |
| Returned To PI Date March 30, 2020 Action Date |
| Returned To PI Date March 30, 2020 |
| Returned To PI Date March 30, 2020 Action Date |
| Returned To PI Date March 30, 2020 Action Date March 30, 2020 |
| Returned To PI Date March 30, 2020 Action Date March 30, 2020 |
| Returned To PI Date March 30, 2020 Action Date March 30, 2020 Comments |
| Returned To PI Date March 30, 2020 Action Date March 30, 2020 Comments Updated By pattonle |
| Returned To PI Date March 30, 2020 Action Date March 30, 2020 Comments Updated By pattonle Update Time |
| Returned To PI Date March 30, 2020 Action Date March 30, 2020 Comments Updated By pattonle |

| Description Submitted to IRB Date March 23, 2020 Action Date March 23, 2020 Comments Submitted to IRB Updated By Szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments Protocol created | |
|---|---|
| Date March 23, 2020 Action Date March 23, 2020 Comments Submitted to IRB Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | Submitted to IRB |
| March 23, 2020 Action Date March 23, 2020 Comments Submitted to IRB Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | |
| Action Date March 23, 2020 Comments Submitted to IRB Updated By SZVONAr Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | Date |
| March 23, 2020 Comments Submitted to IRB Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | March 23, 2020 |
| Comments Submitted to IRB Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | Action Date |
| Submitted to IRB Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | March 23, 2020 |
| Submitted to IRB Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | Comments |
| Updated By szvonar Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | |
| Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | |
| Update Time 2020-03-23T12:00:00.000Z Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | |
| Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | szvonar |
| Description Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | Update Time |
| Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | 2020-03-23T12:00:00.000Z |
| Protocol Created Date January 24, 2020 Action Date January 24, 2020 Comments | Description |
| Date January 24, 2020 Action Date January 24, 2020 Comments | |
| January 24, 2020 Action Date January 24, 2020 Comments | |
| Action Date January 24, 2020 Comments | Date |
| January 24, 2020 Comments | January 24, 2020 |
| Comments | January 24, 2020 |
| Protocol created | Action Date |
| I | Action Date January 24, 2020 |
| Updated By | Action Date January 24, 2020 Comments |
| szvonar | Action Date January 24, 2020 Comments Protocol created |
| | Action Date January 24, 2020 Comments Protocol created Updated By |

Update Time

2020-01-24T12:00:00.000Z

#### **Administrative Details Form**

Protocol Details

9031
Protocol Type
Expedited

Billing Account #

Study Status

#### **Submission Details**

9000

**Submission Review Level** 

Expedited

9030

**Expedited Category.** 

Category 5: Data or specimens that have been or will be collected for nonresearch purposes

Category 6: Data from voice, digital, or image recordings

Category 7: Survey, interview, focus groups, human factor, group behavior or characteristics

9002

Criteria for Approval. Select to confirm.

Approved: The criteria for approval of the research are satisfied in accordance with IU HRPP Policies, and applicable federal regulations.

| Protocol Determinations |
|---|
| 9003 |
| Protocol Level of Risk.<br>Minimal risk |
| 9020 |
| Is renewal required for this research? No |
| 9004 |
| Check all determinations that need to be made. Certificate of Confidentiality |
| 9025 |
| Certificate of Confidentiality. The research is subject to the NIH Policy for Issuing Certificates of Confidentiality and therefore has been issued a Certificate. |
| 9028 |
| Other Determinations. |